CLINICAL TRIAL: NCT00703573
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Efficacy and Safety Study of 2 Doses of S-777469 (400 mg BID and 800 mg BID) in Patients With Atopic Dermatitis
Brief Title: A Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of 2 Doses of S-777469 in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0721D1424
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — S-777469

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): S-777469 400 mg BID (two 200 mg tablets of S-777469 and two tablets of placebo BID)
  Interventions: Drug: S-777469 400 mg; Drug: Placebo
- Group B (Experimental): S-777469 800 mg BID (four 200 mg tablets of S-777469 BID)
  Interventions: Drug: S-777469 800 mg
- Group C (Placebo Comparator): Placebo BID (four tablets of placebo BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-777469 400 mg — S-777469 400 mg BID
  Arms: Group A
Drug: S-777469 800 mg — S-777469 800 mg BID
  Arms: Group B
Drug: Placebo — Placebo BID
  Arms: Group A; Group C

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 2 doses of S-777469 in patients with atopic dermatitis.

ELIGIBILITY:
Screening Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be screened and enrolled into the single-blind period:

* Males or females between 18 and 65 years of age at the time of obtaining the written informed consent
* Patient understands the study procedures and agrees to participate in the study by giving written informed consent
* Patient agrees to allow digital photographs of atopic dermatitis (AD)-affected target areas during the study
* Patient satisfies the diagnostic criteria for AD as defined by the criteria of Hanifin and Rajka (Acta Derm Venereol.1980;92[suppl]:44-47; J Am Acad Dermatol.2003;49[6]:1088-1095), as follows:

Must have 3 or more basic features:

* Pruritis
* Typical morphology and distribution: flexural lichenification or linearity
* Chronic or chronically relapsing dermatitis
* Personal or family history of atopy (asthma, allergic rhinitis, atopic dermatitis)

Plus 3 or more minor features:

* Xerosis
* Ichthyosis/palmar hyperlinearity/keratosis pilaris
* Early age of onset
* Tendency toward cutaneous infections (esp. Staphylococcus aureus and Herpes simplex) /impaired cell-mediated immunity
* Tendency toward non-specific hand or foot dermatitis
* Nipple eczema
* Cheilitis
* Recurrent conjunctivitis
* Dennie-Morgan infraorbital fold
* Keratoconus
* Anterior subcapsular cataracts
* Orbital darkening
* Facial pallor/facial erythema
* Pityriasis alba
* Anterior neck folds
* Itch when sweating
* Intolerance to wool and lipid solvents
* Perifollicular accentuation
* Food intolerance
* Course influenced by environmental/emotional factors
* White dermographism/delayed blanch
* Immediate (type I) skin test reactivity (Provide test results within one year of Screening date.)
* Elevated serum IgE.

  * Patient has negative laboratory results for hepatitis B surface antigen and IgG anti- Hepatitis B core, hepatitis C virus antibodies, and human immunodeficiency virus (HIV) antibody tests at screening
  * Serum creatinine and blood urea nitrogen are in the normal range at screening
  * Female patients of child bearing potential must have a negative pregnancy test at screening and Day-14
  * Patient has a negative screen for drugs of abuse at screening
  * Patient does not have a history or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal or urological disease
  * Patient does not have liver function test results >1.25 the upper limit of normal NOTE: Under no circumstances should a patient who did not qualify regarding liver function tests (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST]) be re-screened and/or re-qualified
  * Patient does not have QTc > 450 (males) or > 470 (females) at screening

Randomization Inclusion Criteria:

Patients eligible to be randomized to double-blind treatment must satisfy all of the following inclusion criteria:

* Patient has all of the following at the end of the single-blind period (Day 1, just before randomization to study drug):

  * Physician's Global Assessment (PGA) ≥ 2 but ≤ 4.
  * The average of the scores recorded from the evening of Day -3 to the morning of Day 1 (Baseline value) of the Numerical Rating Scale (NRS) is ≥ 4.
  * The average of the scores recorded from the evening of Day -3 to the morning of Day 1 (Baseline value) of the Behavior Rating Scale (BRS) is ≥ 2
* Patient has negative laboratory results for hepatitis B surface antigen, IgE anti-Hepatitis B core, hepatitis C virus antibodies, and HIV antibody tests at screening
* Female patients of child bearing potential must have a negative pregnancy test at screening, single-blind period (Day-14) and baseline (Day 1)
* Serum creatinine and blood urea nitrogen are in the normal range at screening
* Patient has negative screen for drugs of abuse at screening and single-blind (Day-14)
* Use of adequate birth control by men and women, if of reproductive potential and sexually active. Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 2 weeks after the last dose of study drug

  * For females, adequate birth control methods will be defined as: hormonal contraceptives, intrauterine device or double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam
  * For males adequate birth control methods will be defined as double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam
  * For females, menopause is defined as one year without menses; if in question, a follicle-stimulating hormone of >40 U/ml must be documented. Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable
* Patient has not used any treatments for AD prior to Day 1, using the following time periods:

  * Systemic (inhaled, oral, suppository or immediate release injectable, depot or sustained-release injectable) corticosteroids, cytostatic drugs, or other immunosuppressant drugs: 5 weeks prior to Day 1
  * Topical immunosuppressant drugs: 4 weeks prior to Day 1
  * Phototherapy, specific desensitization therapy, nonspecific disease-modulating therapy and elimination diet therapy: 4 weeks prior to Day 1
  * Any drugs that are known inhibitors or inducers of Cytochrome P450 isozyme cytochrome CYP2C9: 2 weeks prior to Day 1
  * Systemic antibiotics: 4 weeks prior to Day 1
  * Topical steroids or tar preparations: 2 weeks prior to Day 1
  * Antihistamines, histamine-added γ-globulin preparations, desensitization therapy, or other nonspecific disease-modifying therapies: 2 weeks prior to Day 1
  * Herbal preparation, cosmetic or emollient preparations other than those issued during the screening and single-blind periods: 2 weeks prior to Day 1. Use of cosmetic make-up will be allowed
  * Acetaminophen, acetaminophen-containing products, or non-steroidal anti-inflammatories: 2 weeks prior to Day 1
  * Any other investigational drug or device within 8 weeks prior to Day 1
* Patient is willing to completely avoid the use of any prescription or nonprescription treatments for AD , including over-the-counter drugs or any topical preparations, other than those topical emollient preparations provided by the study site during the screening period and thereafter, as needed. Use of hormone replacement therapy (for postmenopausal females) and/or use of hormonal contraceptive(s), intrauterine device, or double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam will be allowed. Use of topical antibiotics will be allowed during the study

Exclusion Criteria:

Patients satisfying any of the following exclusion criteria are not eligible for enrollment into the double-blind treatment period:

* Patient is under the age of legal consent, is mentally or legally incapacitated and/or has significant emotional problems at the time of study entry
* Patient has an active dermatologic condition other than AD which may confound the diagnosis or evaluation of AD, such as scabies, allergic contact dermatitis, seborrheic dermatitis, cutaneous lymphoma, or psoriasis
* Patient has a history of malignancy not in remission for >5 years, with the exception of cutaneous basal cell carcinoma and cutaneous squamous cell carcinoma
* Presence of comorbid conditions that would preclude participation in the study, including:

  * Immune compromised state, including recent chemotherapy, immunotherapy, or organ transplant
  * History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal or urological disease
  * Signs and symptoms of eczema herpeticum within the preceding 12 months or cellulitis within preceding 3 months
  * Positive results for HIV infection at screening
  * History or clinical manifestations of significant neurological (e.g., epilepsy) or psychiatric disorders (e.g., history of suicide attempt; history of psychiatric episodes resulting in hospitalization)
  * An active intercurrent infection
  * History of clinically significant hypersensitivity, anaphylaxis, or allergies to any drug compound, which resulted in a severe adverse event
  * Liver function tests (ALT, AST) >1.25 times the upper limit of normal at Screening. (refer to Covance Lab Manual for reference ranges) Note: Under no circumstances should a patient who did not qualify regarding liver function tests (ALT and/or AST) be re-screened and/or re-qualified
* Patient has any acute or chronic condition or prior therapy that, in the opinion of the Investigator, would limit the patient's ability to complete and/or participate in this clinical study or otherwise would make the patient unsuitable for this study
* Patient has a history of drug abuse within 1 year prior to Day 1
* Patient consumes excess amounts of alcohol, defined as exceeding an average of 14 drinks/week (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor, or any combination of them) within 2 months prior to Day -14 (beginning of single-blind period) or is unwilling to comply with the restricted use of alcohol (as defined above, no more than 14 drinks/week) from screening, throughout the study, and until study completion (follow-up visit).
* Patient uses any prohibited concomitant medications at any time during the study
* Patient is pregnant or lactating or intends to become pregnant or, in the case of a male patient, intends to father a child during the study period and for 2 weeks after the last dose of study medication
* Patient has poor peripheral venous access that may limit blood sampling for clinical laboratory or pharmacokinetic analysis
* Patient has participated in any other investigational study drug or device trial in which receipt of an investigational study drug or device occurred within 8 weeks prior to Day 1
* Prior exposure to S-777469
* Any reason which, in the opinion of the Investigator, interferes with the ability of the patient to participate in or complete the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of S-777469 was assessed by Physician's Global Assessment (PGA) and Numerical Rating Scale (NRS) | Change from baseline to 12 weeks
  Physician's Global Assessment
Safety was assessed by repeated clinical evaluation and evaluation of treatment-emergent adverse events. It included vital signs, medical history, concomitant medications, physical examination, 12-lead ECGs, and standard clinical laboratory safety tests | Baseline to 12 weeks
  Safety, determined by Adverse event frequency and changes in laboratory values

SECONDARY OUTCOMES:
Efficacy was assessed by PGA, NRS, Behavioral Rating Scale, Eczema Area and Severity Index Score, Investigator panel treatment-blind comparative review ratings of digital photography of affected areas, and Thymus and Activation-Regulated Chemokine | Changes from baseline to various pre-defined time-points during the 12 week study
  Assessment of PGA, NRS, Behavioral Rating Scale, Eczema Area and Severity Index Score, Investigator panel treatment-blind comparative review ratings of digital photography of affected areas, and Thymus and Activation-Regulated Chemokine
Pharmacokinetic analysis of the concentration of unchanged parent drug (S-777469) in trough samples | From Baseline during Week 1
  The concentration of S-777469 will be evaluated to determine when steady state is achieved

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (31):
- United States (31):
  - Hot Springs, Arkansas
  - Los Angeles, California
  - Oceanside, California
  - Riverside, California
  - Denver, Colorado
  - Coral Gables, Florida
  - West Palm Beach, Florida
  - Alpharetta, Georgia
  - Boise, Idaho
  - Arlington Heights, Illinois
  - Evansville, Indiana
  - South Bend, Indiana
  - Fridley, Minnesota
  - Omaha, Nebraska
  - Berlin, New Jersey
  - Paramus, New Jersey
  - Stony Brook, New York
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Johnston, Rhode Island
  - Goodlettsville, Tennessee
  - Knoxville, Tennessee
  - Austin, Texas
  - College Station, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - West Jordan, Utah
  - Lynchburg, Virginia
  - Norfolk, Virginia